CLINICAL TRIAL: NCT04699929
Title: A Open-Label, Phase I Dose Escalation Study to Evaluate the Safety, Tolerability,Efficacy and Pharmacokinetics of YH001 in Subjects With Advanced Solid Tumors
Brief Title: A Study to Evaluate YH001 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH001003
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-05

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/treatment (Experimental): All subject will receive YH001 intravenously as single agent every three weeks (Q3W) for up to 1 years, until intolerable toxicity, confirmed disease progression, withdrawal of consent, or Investigator decision, whichever comes first.
  Interventions: Drug: YH001

INTERVENTIONS:
Drug: YH001 — YH001 will be administered intravenously over 60minutes every three weeks (Q3W) for up to 1 years .

SUMMARY:
This is an open-label, dose-escalation study of the study drug YH001 . The study is designed to determine the safety, tolerability and maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of YH001 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a single arm clinical trial in subjects with advanced solid tumor receiving multiple doses of YH001 intravenously (IV). YH001 will be administered (IV) in 19-37 patients with advanced solid tumors. An accelerated titration method followed by a traditional 3+3 dose escalation scheme will be utilized to determine MTD(maximum tolerated dose) and/or RP2D(recommended phase 2 dose). Patients will be dosed at Dose A, Dose B, Dose C, Dose D, Dose E, Dose F and Dose G every 3 weeks (Q3W) for 15 weeks (5 cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 18 years;
2. Patients with histologically or cytologically confirmed solid tumors who have failed standard of care or have no standard of care;
3. Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1;
4. Have life expectancy of at least 3 months based on investigator's judgement;
5. Organ function levels must meet the following requirements:

   A:Hematology: absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelet count ≥ 100 x 10^9/L, hemoglobin (Hb) ≥ 100 g/L ; B:Liver: serum total bilirubin (TBIL) ≤ 1.5 × the upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN (patients with primary liver cancer or liver metastases: AST and/or ALT < 5 × ULN); C:Kidney: creatinine clearance (CrCL) ≥ 50 mL/min;
6. International normalized ratio (INR) ≤ 1.5 × ULN, prothrombin time (PT) ≤ 1.5 × ULN, activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN;
7. All women of reproductive potential, men whose partner is a woman of reproductive potential, or their spouses should use adequate barrier contraception throughout the study and for 3 months after the last dose;
8. Voluntary and agree to sign the informed consent and follow the study treatment protocol as well as follow-up plan.

Exclusion Criteria:

1. Subjects with prior anti-CTLA-4 checkpoint inhibitors should be excluded;
2. Patients with any other malignancy within the past 5 years or currently, except for completely cured non-melanoma skin cancer, carcinoma in situ of the cervix, and ductal carcinoma in situ of the breast;
3. Received other anti-tumor therapies (such as chemotherapy, radiotherapy, surgery, endocrine therapy, targeted therapy, immunotherapy, etc.) within 4 weeks or 5 half-lives (whichever is longer) before the first dose, or received modern Chinese medicine preparations with anti-tumor effect approved by NMPA within 2 weeks prior to the first dose;
4. Major surgery (excluding vascular access establishment surgery) was received within 4 weeks prior to the first dose;
5. Has received immunosuppressive therapy within 4 weeks prior to the first dose. However, enrollment is permitted under the following circumstances:
6. In the absence of active autoimmune disease, patients are allowed to receive inhaled or topical glucocorticoids, or other glucocorticoids at doses ≤ 10 mg/day prednisone equivalent.

   Patients with primary central nervous system (CNS) tumors, or symptomatic CNS tumors, or spinal cord compression, or carcinomatous meningitis; with the following exceptions:

   Patients with asymptomatic brain metastases (i.e., no progressive central nervous system symptoms due to brain metastatic sites, no need for corticosteroids, and lesion size ≤ 1.5 cm); Patients whose symptoms are controlled by treatment, i.e., their condition is stable and asymptomatic at least 4 weeks after treatment;
7. Use of any other study drug within 4 weeks prior to the first dose, or participation in other clinical studies;
8. Have received live or attenuated vaccines within 4 weeks prior to the first dose;
9. Patients with known severe allergic reactions (≥ Grade 3) to the active ingredient and excipients of the investigational drug, other monoclonal antibodies or "Immuno-oncology drugs;
10. Toxic and side effects caused by prior anti-tumor therapy before the first dose did not recover to ≤ Grade 1 (CTCAE v5.0), except for alopecia and sensory neuropathy below Grade 2;
11. History of interstitial pneumonia or non-infectious pneumonitis requiring corticosteroids, except for radiation therapy, or current presence of interstitial pneumonia or non-infectious pneumonitis;
12. ≥ Grade 2 immune-related pneumonitis occurred during prior immunotherapy;
13. History of ≥ Grade 3 immune-related adverse reactions or any adverse reactions leading to discontinuation of immunotherapy during prior immunotherapy;
14. Past or existing active tuberculosis ;
15. Patients with active auto-immune disease, history of auto-immune disease requiring systemic therapy, or history of auto-immune disease within 2 years prior to the first dose, with the following exceptions: leucoderma, childhood asthma/specific reactions, type I diabetes mellitus, hypothyroidism which can be treated with replacement therapy;
16. Clinically uncontrollable disease, including, but not limited to, severe diabetes (fasting glucose > 250 mg/dl,1 mg/dl = 18 mmol/L), uncontrollable hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg), or other serious disease requiring systemic treatment;
17. Patients with active infections, including active hepatitis B, active hepatitis C, and human immunodeficiency virus infection;
18. Patients with active infection requiring intravenous infusion;
19. Serious cardiovascular and cerebrovascular diseases, such as cerebrovascular rupture, stroke, myocardial infarction, unstable angina pectoris, congestive heart failure (New York Heart Association Grade ≥ II), severe uncontrolled arrhythmia, etc., occurred within 6 months prior to the first dose;
20. Patients with clinically significant ECG abnormalities: QTcF ≥ 470 msec (corrected by Fridericia), or having history of congenital long QT syndrome, or taking any known QTc prolonging medication;
21. Patients who have received allogeneic bone marrow transplant or organ transplant;
22. Known psychiatric disorders, drug abuse, drug use, or alcohol dependence that may affect trial compliance;
23. Other conditions that were considered not suitable for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-10-08 (Actual); Study Completion 2022-10-08 (Actual)

PRIMARY OUTCOMES:
Overall safety and tolerability profile of YH001 (adverse events) | From screening up to 1 year
  The safety profile of YH001 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Maximum tolerated dose (MTD) | Cycle 1 of each cohort. Duration of one cycle is 21 day
  The MTD will be determined based on the data of safety and tolerability
Recommended phase 2 dose (RP2D) | Cycle 1 of each cohort. Duration of one cycle is 21 day
  The RP2D will be determined based on the data of safety and tolerability

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) | Up to 1 year
  To determine the PK profile of YH001
Trough concentration before the next dose is administered (Ctrough) | Up to 1 year
  To determine the PK profile of YH001
Time to reach maximum serum concentration (Tmax) | Up to 1 year
  To determine the PK profile of YH001
Clearance (CL) | Up to 1 year
  To determine the PK profile of YH001

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital,Sichuan University, Chengdu, Sichuan